CLINICAL TRIAL: NCT00705328
Title: Families First Edmonton: The Comparative Effects and Expense of Four Models of Augmenting Services for Low-income Families
Brief Title: Families First Edmonton (FFE)
Acronym: FFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Maria Mayan, Vice Provost - Health Sciences Council; Professor - Nursing, University of Alberta
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 137444
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Low-Income Population
Keywords: low-income families; children; recreation; family healthy lifestyle; linkages to community resources; Families with low incomes; working poor; welfare recipients

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Primary Health Care Model (PRMHLTH)
- 2 (Experimental)
  Interventions: Behavioral: Recreation Coordination Model (REC)
- 3 (Experimental)
  Interventions: Behavioral: Comprehensive Model (COMP)

INTERVENTIONS:
Behavioral: Primary Health Care Model (PRMHLTH) — Primary health care service delivery
  Arms: 1
Behavioral: Recreation Coordination Model (REC) — Recreation coordination service delivery
  Arms: 2
Behavioral: Comprehensive Model (COMP) — a comprehensive service delivery model consisting of PRMHLTH plus REC.
  Arms: 3

SUMMARY:
This study is designed to provide clear evidence for health and social policymakers about the influence of alternate service-delivery models and practices on enhancing and sustaining low-income family linkages to available services. A challenge faced by Canadian health and social service providers is to promote health for low-income families in a proactive and cost-effective manner. Families with low incomes experience an array of health and social barriers that compromise their resilience, lead to negative family outcomes, and act as barriers to available services. Family barriers are compounded by service delivery barriers and result in reduced opportunities for effective, primary-level services and in increased use of secondary-level services (e.g., emergency room visits, emergency intervention, police involvement), with the obvious increase in costs. Randomized-controlled trials are rare in community-based intervention research.

This Families First Edmonton randomized-controlled trial (RCT) will enable testing of innovative service-delivery models and provide an opportunity for evidence-based decision making for Canadian policy makers. Critical information will be provided about

1. optimizing cost effectiveness for public systems
2. the long-term effects on the health of low-income family members
3. mechanisms that intervene between the interventions and their effect on the health of low-income family members
4. building on previous research and on community-based initiatives
5. promoting knowledge transfer

ELIGIBILITY:
Inclusion Criteria:

* Participant families will

  1. have received low-income assistance either in the form of

     1. Alberta Works Income Support
     2. Alberta Child Health Benefits,
     3. Alberta Works Adult Health Benefits
     4. participating in City of Edmonton Leisure Access Program
     5. living in Capital Region Housing
  2. have a child or children between 0 and 12 years of age
  3. reside in city of Edmonton
  4. be able to provide signed consent

Exclusion Criteria:

* Potential study participants will be excluded if they refuse to give informed consent to be interviewed
* are unable to read and write English and an appropriate translator is not available
* have plans to move outside the region
* are unwilling to participate for the entire follow-up period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2005-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Increased linkages between low income families and established services in their communities | Baseline, 12-month, 24-month, 36-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jane Drummond, PhD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Human Resources and Employment, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Browne G, Byrne C, Roberts J, Gafni A, Whittaker S. When the bough breaks: provider-initiated comprehensive care is more effective and less expensive for sole-support parents on social assistance. Soc Sci Med. 2001 Dec;53(12):1697-710. doi: 10.1016/s0277-9536(00)00455-x. PMID 11762894
- [Derived] Drummond J, Wiebe N, So S, Schnirner L, Bisanz J, Williamson DL, Mayan M, Templeton L, Fassbender K; Community-University Partnership for the Study of Children, Youth, and Families. Service-integration approaches for families with low income: a Families First Edmonton, community-based, randomized, controlled trial. Trials. 2016 Jul 22;17:343. doi: 10.1186/s13063-016-1444-8. PMID 27449358
- [Derived] Drummond J, Schnirer L, So S, Mayan M, Williamson DL, Bisanz J, Fassbender K, Wiebe N. The protocol for the Families First Edmonton trial (FFE): a randomized community-based trial to compare four service integration approaches for families with low-income. BMC Health Serv Res. 2014 May 19;14:223. doi: 10.1186/1472-6963-14-223. PMID 24885729